CLINICAL TRIAL: NCT00984672
Title: Prospective Evaluation of Radiculitis Following Use of Bone Morphogenetic Protein-2 for Interbody Arthrodesis in Spinal Surgery
Brief Title: Evaluation of Radiculitis Following Use of Bone Morphogenetic Protein-2 for Interbody Arthrodesis in Spinal Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ahmad Nassr, PI, Mayo Clinic
Other Study IDs: 08-008802
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Lumbar Degenerative Disease
Keywords: Lumbar Degenerative Disease; Bone Morphogenetic Protein; TLIF

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bone morphogenetic protein within an interbody cage: Transforaminal Lumbar Interbody Fusion with the use of BMP
- Other bone grafting techniques within cage (non-BMP): Use of iliac crest autograft, allograft, or local autogenous bone grafting within the cage during Transforaminal Lumbar Interbody Fusion.

SUMMARY:
Clinician directed use of bone morphogenetic proteins (BMPs) in ways other than FDA approved, has increased recently due to the morbidity associated with harvest of iliac crest bone graft in spinal arthrodesis procedures. FDA approved for the use in anterior lumbar fusions with LT Cage, other clinical applications of these proteins is becoming widely adopted due to their effectiveness in forming bone and facilitating fusion. Clinicians have realized while these proteins are potent stimulators of bone formation there have been anecdotal reports of increased rates of radicular pain in the postoperative period when used in interbody arthrodesis procedures. Speculation as to the mechanism of this radiculitis is postulated to be due to the inflammatory effects of these proteins. Excess bone overgrowth around the spinal nerves in proximity to the fusion cage has been reported. No prospective studies have been performed assessing the incidence and etiology of this complication. The investigators propose a prospective study evaluating the incidence of this complication as well as postoperative imaging studies to help determine whether bony overgrowth is indeed occurring adjacent to the effected spinal nerves.

ELIGIBILITY:
Inclusion Criteria:

* male or female age 18-75
* candidate for TLIF
* Lumbar levels L1-S1

Exclusion Criteria:

* more than 3 TLIF levels
* had a previous fusion attempt at involved level(s)
* had more than 2 previous open, lumbar spine procedures at the involved level(s)
* currently implanted with anterior instrumentation at the involved level(s)
* BMI >40
* active localized or systemic infection
* presence of a disease entity or condition which significantly affects the possibility of bony fusion
* has immunosuppressive disorder actively requiring treatment
* pregnant or interested in becoming pregnant during the study
* has a known sensitivity to device materials
* mentally incompetent or is a prisoner
* currently a participant in another study for the same indications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18-75 with lumbar degenerative conditions including degenerative disk disease, spondylolisthesis with significant back and or leg complaints that have failed greater than 6 weeks of conservative therapy that are felt to be candidates for posterior lumbar instrumented fusion with transforaminal interbody fusion (TLIF).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2009-03; Primary Completion 2016-04-21 (Actual); Study Completion 2016-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Nassr, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials